CLINICAL TRIAL: NCT04459988
Title: Enhanced Regulatory Functions of Bregs With Ocrelizumab in Multiple Sclerosis
Brief Title: Mechanistic Study of Ocrevus
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David A. Fox, MD, Professor of Rheumatology and Internal Medicine, University of Michigan
Other Study IDs: HUM00066792
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Ocrevus; B cell; T cell; cytokines
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be collected after 3, 6, 9, 12, 18 and 24 months of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with MS: Patients with MS who have been newly prescribed Ocrevus
  Interventions: Drug: Ocrelizumab
- Healthy Controls: Healthy Controls

INTERVENTIONS:
Drug: Ocrelizumab — Description Needed
  Other Names: Ocrevus
  Groups: Patients with MS

SUMMARY:
The purpose of this study is to investigate the immune cell and other factor changes with Ocrevus in Multiple Sclerosis (MS) patients. Researchers will recruit 35 participants for this study. Patients will be enrolled from the Multiple Sclerosis Center at the University of Michigan Health System in Ann Arbor. The goal of the study is to understand the role of regulatory B cell, T cell and other factors in mediating the therapeutic effects of Ocrevus.

ELIGIBILITY:
Inclusion Criteria:

Patients with MS either with relapsing or primary progressive course; who are newly starting on ocrelizumab (Ocrevus) at the time of enrollment

OR

Healthy controls who do not have a significant medical conditions such as cancer, chronic infection, or autoimmune disease, have not taken steroids in the past 2 months, and who are not on an immune suppressant medication.

* Ability to give informed consent
* Willing to have blood drawn as scheduled in the protocol
* Willing and able to complete all procedures and evaluations related to the study

Exclusion Criteria:

* Medical or psychiatric conditions that may affect the patient's ability to give informed consent
* Has received an experimental drug within 30 days of enrollment
* Concomitant other disease modifying medications (such as Rebif, Betaseron, Avonex, Copaxone, Gilenya, Tecfidera, Aubagio, Mayzent, Mavenclad, Alemtuzumab, methotrexate, azathioprine, Novantrone, cyclophosphamide, cyclosporine, Tysabri, Rituxan, Ocrevus, etc.)
* Has any contraindication to high-dose immunotherapy, including pregnancy, trying to become pregnant, or breast feeding during the study
* Active hepatitis B virus infection
* History of life-threatening infusion reaction to Rituxan or Ocrevus
* Chronic infection or any severe acute infection within 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit 25 MS patients (Group 1; include 5-10 PPMS and 15-20 RRMS). Meanwhile, 10 healthy controls (Group 2; HCs) will be recruited to establish baseline immune cell profiles. The patients and healthy controls will be recruited at the University of Michigan Neurology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Change in frequency of regulatory B cells | From baseline to 24 months
  Percentage B cells measured by flow cytometry. Compare Ocrevus treatment to baseline and to healthy controls

SECONDARY OUTCOMES:
Change in frequency of T cell subtypes | From baseline to 24 months
  Percentage of T cells measured by flow cytometry. Compare Ocrevus treatment to baseline and to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mao-Draayer, MD/PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No